CLINICAL TRIAL: NCT04818021
Title: Contribution of the Somatosensory System to Speech Perceptual Processing Aim 3
Brief Title: Contribution of the Somatosensory System to Speech Perceptual Processing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of funding
Sponsor: Yale University (Other)
Collaborators: McGill University (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000025475_b; R01DC017439 (NIH)
Record Dates: First submitted 2021-03-19; First posted 2021-03-26 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Speech; Consolidation
MeSH Terms: conditions — Speech | interventions — Acclimatization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adaptation to Altered Auditory Feedback (Experimental): Adaptation to Altered Auditory Feedback
  Interventions: Behavioral: Adaptation
- Adaptation to Altered Auditory Feedback + Forward Skin Stretch (Experimental): Adaptation to Altered Auditory Feedback + Forward Skin Stretch
  Interventions: Behavioral: Adaptation; Behavioral: Facial Skin Stretch
- Adaptation to Altered Auditory Feedback + Backward Skin Stretch (Experimental): Adaptation to Altered Auditory Feedback + Backward Skin Stretch
  Interventions: Behavioral: Adaptation; Behavioral: Facial Skin Stretch
- Speech Repetition Control (Experimental): Speech Repetition Control
  Interventions: Behavioral: Adaptation

INTERVENTIONS:
Behavioral: Adaptation — Sensorimotor adaptation in speech
Behavioral: Facial Skin Stretch — Facial skin stretch
  Arms: Adaptation to Altered Auditory Feedback + Backward Skin Stretch; Adaptation to Altered Auditory Feedback + Forward Skin Stretch

SUMMARY:
These studies test the hypothesis that the repeated pairing of somatosensory inputs with speech sounds, such as occurs during speech motor learning, results in changes to the perceptual classification of speech sounds.

DETAILED DESCRIPTION:
This study will assess changes to the perceptual classification of speech sounds that are related to repeated pairing of somatosensory and auditory inputs (as would occur during speech motor learning). Before and after the training, base-line and post-training auditory perceptual performance will be examined in the absence of somatosensory stimulation, in order to evaluate the effects of the pairing on speech perception. Perceptual classification and speech motor learning will both be assessed on a 0 to 100 scale.

ELIGIBILITY:
Inclusion Criteria:

* right handed adults
* no known physical or neurological abnormalities

Exclusion Criteria:

* patients with:
* cardiac pacemaker
* surgical clips or values on the heart
* implants
* metal or metallic fragments in any part of the body
* pregnancy
* claustrophobia
* a personal or family history of epilepsy
* currently taking antipsychotic drugs
* currently taking antidepressant drugs
* currently taking antianxiety drugs.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Speech Motor Learning | Performance as measured at the end of learning (30 minute session)
  Learning is assessed as the change in speech sounds (speech formant frequencies) on a 0 to 100 scale.
Speech Perception | Perception is evaluated prior to and after perceptual training (30 minute session)
  Auditory speech perception evaluates auditory classification and is assessed on a 0 to 100 scale. All conditions of skin stretch involve the same speech perception task.

CONTACTS AND LOCATIONS:
Overall Officials: David Ostry, Principal Investigator — Haskins Laboratories
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2019-04-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT04818021/Prot_001.pdf
  • Informed Consent Form (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT04818021/ICF_000.pdf